CLINICAL TRIAL: NCT02543372
Title: Internet-Delivered Treatments for Pathological Gambling: a Randomized Controlled Trial Comparing the Effects of Added Involvement By Concerned Significant Others
Brief Title: RCT of Internet-Delivered CBT Treatments for Pathological Gambling: Comparing the Effects of Added Involvement From CSOs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm University (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Clara Hellner Gumpert, MD/PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/175-31/5
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Gambling
Keywords: concerned significant other; problem gambling; internet-delivered cognitive-behavioral therapy; behavioral couples therapy
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy

ARMS (2):
- Behavioral Couples Therapy (Experimental): The participants receive 10 modules each containing treatment focusing on gambling and relationship functioning. The modules consist of text, videos, images and assignments. The participants receive support from an assigned therapist via email and telephone. Both the gamblers and the CSOs receive 10 modules each.
  Interventions: Behavioral: Behavioral Couples Therapy (BCT)
- Cognitive Behavioral Therapy (Active Comparator): The participants receive 10 modules each containing treatment focusing on gambling and relationship functioning. The modules consist of text, videos, images and assignments. The participants receive support from an assigned therapist via email and telephone. The gamblers receive 10 modules, but the CSOs do not receive any modules.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Behavioral Couples Therapy (BCT) — BCT integrates cognitive behavioral techniques targeting problem gambling with a large focus on interventions for relationship functioning. The BCT condition requires active participation from both the gambler and the CSO.
  Arms: Behavioral Couples Therapy
Behavioral: Cognitive Behavioral Therapy (CBT) — The CBT integrates cognitive behavioral techniques targeting problem gambling with some interventions for relationship functioning.The CBT condition requires active participation from the gambler, but not for the CSO.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Background: Problem gambling is a public health concern with prevalence rates at 2 %. Problem gambling also severely affects concerned significant others (CSOs). Several studies have investigated the effects of individual treatments based on cognitive behavior therapy (CBT), but there is a shortage in studies on the effect of involving CSOs in treatment. This study aims to compare an intervention based on behavioral couples therapy (BCT) involving a CSO with an individual CBT treatment to determine their relative efficacy. BCT has shown promising results in working with substance abuse, but this is the first time it is used as an intervention for problem gambling. Both interventions will be Internet-delivered and participants will receive e-mail and telephone support.

Method/Design: A sample of at least 100 couples will be randomized to either the BCT condition or the CBT condition. The participants will work through 10 modules over 12 weeks in a secure online environment, and receive support via email and over telephone. Repeated measures will be conducted weekly and at 3, 6 and 12 months follow-up. The primary outcome measure is gambling behavior, defined as time spent and money lost on gambling, as measured by timeline follow-back. Secondary outcomes include gambling related harm, alcohol consumption, relationship satisfaction and mental health for the gambler as well as for the CSO.

Hypotheses: The investigators hypothesize that a) BCT will yield greater reductions on gambling measures than CBT, b) BCT will yield a lower drop-out rate compared to CBT, c) BCT will be superior to CBT on increasing relationship satisfaction, d) relationship functioning will mediate change in gambling behavior in the BCT group and e) reduction in gambling behavior will mediate change in relationship functioning in the CBT group.

ELIGIBILITY:
Inclusion Criteria:

* The CSO is a parent, child, sibling, friend or partner of the gambler.
* Participants are at least 18 years old.
* The gambler is a problem gambler according to Problem Gambling Severity Index.
* Participants must have had a relationship with the gambler for at least 3 months.
* Participants must be able to read and answer questions in Swedish, and is willing to be in contact with a counselor each week.
* Participants must have access to internet.

Exclusion Criteria:

* Participants are currently in any other treatment related to problem gambling.
* The CSO is a problem gambler according to Problem Gambling Severity Index.
* Participants displaying symptoms of severe psychiatric disorders, such as psychotic- or bipolar disorders, judged to require further treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Gambling-Timelime Follow-Back (G-TLFB) | Change from baseline at: [1] weekly during treatment;[2] end of treatment period; follow-ups at [3] month 6 and [4] month 12 after the treatment period.
  Measures money and time spent on gambling by the gambler, as rated individually by the gambler and the CSO.
National Opinion Research Center DSM-IV Screen for Gambling Problems (NODS) | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  Measures consequences of gambling, as rated by the problem gambler.

SECONDARY OUTCOMES:
9-item Patient Health Questionnaire (PHQ-9) | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  Screening for depressive symptoms, as rated individually by the gambler and the CSO.
The Generalized Anxiety Disorder 7-item (GAD-7) | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  Screening for anxiety, as rated individually by the gambler and the CSO.
Relationship Assessment Scale (generic version) (RAS-G) | Change from baseline at: [1] weekly during treatment;[2] end of treatment period; follow-ups at [3] month 6 and [4] month 12 after the treatment period.
  Measures relationship satisfaction, as rated individually by the gambler and the CSO.
Inventory of Consequences Scale for the Gambler and CSO | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  Measures consequences of gambling, as rated individually by the gambler and the CSO.
The Alcohol Use Disorders Identification Test (AUDIT) | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  Measures alcohol consumption, as rated individually by the gambler and the CSO.
Dissociative Experiences while Gambling | Change from baseline at: [1] end of treatment period; follow-ups at [2] month 6 and [3] month 12 after the treatment period.
  Measures dissociative experiences while gambling, as rated by the gambler.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Hellner Gumpert, MD/PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Nilsson A, Magnusson K, Carlbring P, Andersson G, Hellner Gumpert C. Effects of added involvement from concerned significant others in internet-delivered CBT treatments for problem gambling: study protocol for a randomised controlled trial. BMJ Open. 2016 Sep 26;6(9):e011974. doi: 10.1136/bmjopen-2016-011974. PMID 27670519
- See also: Public website to convey study information and recruitment — http://www.spelfri.se